CLINICAL TRIAL: NCT02005627
Title: Randomised Placebo-controlled Study of Grass Pollen Allergen Immunotherapy Tablet (AIT) for Seasonal Rhinitis: Time Course of Nasal, Cutaneous and Immunological Outcomes
Brief Title: Grass Pollen Allergen Immunotherapy Tablet (AIT) Time Course Study
Acronym: Pollen+
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: King's College London (Other); ALK-Abelló A/S (Industry); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13IC0847; 2013-003732-72 (EudraCT Number); 13/EM/0351 (Other: United Kingdom (UK) Research Ethics Committee)
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Allergic Rhinitis
Keywords: grass pollen allergy; hayfever; atopy; allergic rhinitis; sublingual immunotherapy tablets
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Grazax; Desensitization, Immunologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grazax (Active Comparator): The active treatment arm will receive active grass pollen immunotherapy tablet (AIT), Grazax Oral Lyophilisate 75,000 standardised quality units tablet (SQ-T) once daily.
  Interventions: Drug: Grazax
- Grazax Placebo (Placebo Comparator): This arm will receive Grazax placebo once daily which contains the same composition as in the active Grazax tablet with the only difference being the exclusion of the grass pollen allergen extract.
  Interventions: Drug: Grazax Placebo

INTERVENTIONS:
Drug: Grazax — The active treatment arm will receive active grass pollen immunotherapy tablet (AIT), Grazax Oral Lyophilisate 75,000 SQ-T once daily.
  Other Names: Grazax 75,000 SQ-T oral lyophilisate; Allergen Immunotherapy Tablet; SQ Standardized Grass Allergy Immunotherapy
  Arms: Grazax
Drug: Grazax Placebo — This arm will receive Grazax placebo once daily which contains the same composition as in the active Grazax tablet with the only difference being the exclusion of the grass pollen allergen extract.
  Other Names: Grazax Placebo tablet
  Arms: Grazax Placebo

SUMMARY:
About 45 million people in Europe have allergic rhinitis (hay fever) - inflammation of the nasal passages causing sneezing, runny nose, nasal congestion, itching and tearing of the eyes. In the United Kingdom (UK), seasonal hay fever due to grass pollen allergy accounts for approximately 7 times more doctors' appointments than asthma. The standard treatment for hay fever consists of treating the symptoms with a nasal spray and an antihistamine. However, in a survey taken in a UK general practice less than 40% of patients with hay fever reported good symptom control with this standard treatment. For those patients with hay fever whose symptoms are not well controlled by treatment with antihistamines and nasal sprays, subcutaneous immunotherapy (SCIT) - (monthly injections of a grass allergen extract for a period of 3-5 years) is an effective alternative, and is approved in the UK on a named patient basis. More recently, allergen immunotherapy tablets (AITs) have been developed, including grass pollen allergen tablets. These have been shown to be highly effective in the treatment of hay fever, with the additional benefit of being convenient for patients, given that they may be taken at home. Grazax® (manufactured by Allergologisk Laboratorium København (ALK)-Abello, Denmark) has UK and European Union (EU) license for use in the treatment of troublesome grass pollen induced hay fever. The aim of this research is to investigate the effects of the AIT treatment on the immune system over time - which changes are taking place and when in the course of treatment. This will provide insight into the complexities of the development of allergen-specific immune tolerance - how harmful allergic responses against innocuous substances such as grass pollen can be overridden.

DETAILED DESCRIPTION:
The study will be conducted over 44 months. We expect to screen 70 atopic patients in order to enroll up to 50 suitable atopic participants to ensure randomisation of at least 40 atopic participants following their baseline visit. Additionally, we shall recruit 20 healthy, non-atopic volunteers. Individuals with moderate to severe grass pollen hay fever, with or without associated seasonal asthma, will be recruited and screened after the pollen season from September through March 2014. Atopic Participants will undergo baseline assessments in December 2013 to March 2014. All screening assessments will be completed before eligible participants are randomized to active or placebo treatment. Atopic participants will then begin AIT treatment in February-March 2014 and continue treatment for 12 months. All atopic participants will be provided with anti-allergic rescue medications (antihistamine tablets, topical intranasal corticosteroids, and eye-drops) throughout the pollen season. Clinical surrogate endpoint assessments and on specific time Points blood, nasal fluid and nasal brushing sampling, will be performed at baseline (January-March 2014), at 4, 8, 12 and 16 weeks after starting the AIT, and at 6 and at 12 months (January-March 2015) of treatment. Nasal mucosal biopsies will be taken at baseline, during the Peak pollen season, and 12 months of treatment. After 12 months of treatment, unblinding will take place. Those atopic participants receiving active AIT treatment will continue therapy for another 12 months followed by a withdrawal phase of 12 months. Blood samples and nasal biopsies will be taken from these participants again at 24 and at 36 months from the initial start of treatment. Those atopic participants on placebo will be offered 24 months of active treatment after unblinding.

20 healthy, non-atopic participants will also be recruited and studied on a single day before and after nasal challenge at one timepoint at 12 months. They will undergo the same clinical and immunological measurements as for the 46 randomised subjects participating in the clinical trial. The healthy subjects will undergo no therapeutic intervention and serve as controls for the immunological measurements.

The study will receive monitoring by:

* the sponsor, Imperial College London

and audits by:

* Medicines for human use (clinical trials) regulations authority (MHRA)

We will assess the clinical data on paper case report forms and will use Inform as a database in order to verify completeness of data entry.

The Inform database also includes normal ranges of parameters if relevant.

Standard Operating Procedures are in place regarding clinical measures (e.g. nasal allergen challenges, nasal biopsies etc.) as well as data management (e.g. the Trial Master File), reporting of adverse events and data collection. All involved investigators are informed about these procedures and have current Good Clinical Practice (GMC) instructions.

Statistical analysis will be with non-parametric statistics taking into account treatment effect baseline values and visit number. Inclusion of 20 participants per group will give greater than 90% power (p=0.05) to detect a 40% reduction in the early phase response (EPR) after nasal challenge (AUC of the TNSS in the first 60 minutes after challenge, a 40% reduction in the skin late phase response (LPR), and a 50% increase in grass pollen allergen specific immunoglobulin G4 (IgG4) for AIT vs. placebo.

Based on more recent nasal allergen challenge studies (Scadding et al, unpublished data; mean 4.63, standard deviation 1.65 for AUC 0-60 minutes post grass pollen nasal challenge in 14 allergic volunteers), inclusion of 13 patients per group will provide 80% power to detect a 40% reduction in AUC after challenge, whereas inclusion of 22 patients per group will provide 80% power to detect a 30% reduction.

Further based on a recent study (Scadding et al, unpublished data; mean 70.14, standard deviation 14.17 for cross-sectional area in cm2 at 8 hours for skin late phase response to intradermal grass pollen injection), inclusion of 7 participants per group will provide 80% power to detect a 30% reduction, whereas inclusion of 10 participants per group will provide 90% power to detect a 30% reduction.

Intent-to-treat (ITT) sample will be defined as all randomized participants. ITT participants will be analysed with the group to which they were randomized, regardless of the medication actually received. If participants drop out post randomisation, they will be invited to complete study assessments throughout the duration of the trial.

Per-protocol (PP) sample will be defined as ITT sample participants who remain in the study for 12 months and in whom the primary endpoints were assessed. Participants in the PP sample must be compliant with study medication, defined as taking 75% or more of their study medication for the duration of the study. Compliance with study medication will be as assessed by pill count for returned AIT/placebo. Participants in the PP sample will be analysed with the group to which they were randomized. The non-atopics will also be included in the PP sample.

Safety sample (SS) will be defined as all enrolled participants.

Analysis of study data will be conducted to address all objectives of the trial and other interrelationships among all data elements of interest to the investigators and of relevance to the objectives of the study. Primary analysis of treatment effect will be conducted under the intention-to-treat (ITT) principle of eligible patients, whereby outcome data from all eligible patients will be included regardless of treatment compliance. In addition to the analyses described in sections below, summary descriptive statistics will be provided in the following manner: continuous data will be summarized descriptively by mean, standard deviation, median, and range; categorical data will be presented as enumerations and percentages.

Analysis of primary endpoint:

The primary endpoint will be analysed using the ITT and the PP sample. The analysis of the primary endpoint will compare the mean EPR to nasal challenge recorded by the TNSS during the first 60 minutes after the nasal challenge, at 12 months of therapy. Comparison between active and placebo groups will be assessed using ANOVA at the 0.05 level of significance.

Analysis of secondary endpoint:

All secondary analyses will be treated as supportive. P-values will be presented for the secondary endpoints but will not be adjusted for multiplicity and should be interpreted with caution. Findings will be evaluated in the context of the available body of knowledge and with respect to other findings.

ELIGIBILITY:
Atopic Participants:

Inclusion Criteria:

* age 18 to 65
* grass pollen-induced allergic rhinoconjunctivitis for at least 2 years with peak symptoms in May-July.
* moderate to severe rhinoconjunctivitis symptoms with or without mild seasonal asthma interfering with usual daily activities/sleep.
* rhinoconjunctivitis that remains troublesome despite treatment with either antihistamines or nasal corticosteroids during the grass pollen season.
* Positive skin prick test response (wheal diameter ≥ 3 mm) to timothy grass pollen.
* Positive specific immunoglobulin E (IgE), defined as IgE immunoCAP ≥ 0.7 Immuno Solid Phase Allergenchip (ISAC) standardized units (ISU), against timothy grass pollen.
* if applicable a negative urine pregnancy test and willingness to use an effective form of contraception for the duration of involvement in the study.
* The ability to give informed consent and comply with study procedures.
* A positive grass pollen nasal allergen challenge test as defined by a total nasal symptom score (TNSS) of at least 7/12 after 5 minutes with an allergen dose of 5,000 bioequivalent units (BU)/ml.

Exclusion Criteria:

* Previous grass pollen allergen immunotherapy.
* Prebronchodilator forced expiratory volume at one second (FEV1) < 70% of predicted value out of grass-pollen season.
* A clinical history of symptomatic allergic rhinitis and/or asthma caused by an allergen to which the participant is regularly exposed.
* Perennial asthma requiring regular inhaled corticosteroids.
* Seasonal symptoms outside the grass-pollen season.
* History of emergency visit or hospital admission for asthma in the previous 12 months.
* History of chronic obstructive pulmonary disease.
* History of significant recurrent acute sinusitis.
* History of chronic sinusitis.
* At screening visit evidence for upper respiratory tract infection.Participants may be re-evaluated for eligibility after symptoms resolve.
* Current smokers or a history of ≥ 5 pack years.
* History of life-threatening anaphylaxis or angioedema.
* Ongoing systemic immunosuppressive treatment.
* The use of any investigational drug within 30 days of the screening visit.
* The presence of any medical condition that the investigator deems incompatible with participation in the study.
* History of fish allergy with positive skin test and/or positive specific IgE test to vertebrate/finned fish.
* Contraindications taking Grazax.

Non-Atopic:

Inclusion Criteria:

* age 18 to 65.
* Negative skin prick test response to timothy grass pollen and panel of aeroallergens.
* Negative specific IgE, defined as IgE immunoCAP < 0.35 ISU, against timothy grass pollen.
* If applicable a negative urine pregnancy test at the time of screening and willingness to use an effective form of contraception for the duration of involvement in the study.
* The ability to give informed consent and comply with study procedures.

Exclusion criteria:

* Previous grass pollen allergen immunotherapy.
* Prebronchodilator FEV1 < 70% of predicted value out of grass-pollen season.
* symptomatic allergic rhinitis and/or asthma caused by an allergen to which the participant is regularly and perennially exposed (e.g. cat dander).
* Perennial asthma requiring regular inhaled corticosteroids.
* Seasonal symptoms outside or during the grass-pollen season.
* History of emergency visit or hospital admission for asthma in the previous 12 months.
* History of chronic obstructive pulmonary disease.
* History of significant recurrent acute sinusitis.
* History of chronic sinusitis.
* At screening visit, current symptoms of upper respiratory tract infection. Participants may be re-evaluated for eligibility after symptoms resolve.
* Current smokers or a history of ≥ 5 pack years.
* History of life-threatening anaphylaxis or angioedema.
* Ongoing systemic immunosuppressive treatment.
* The use of any investigational drug within 30 days of the screening visit.
* The presence of any medical condition that the investigator deems incompatible with participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Durham, Prof., Principal Investigator — Imperial College London
Locations (1):
- NHS Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steveling EH, Lao-Araya M, Koulias C, Scadding G, Eifan A, James LK, Dumitru A, Penagos M, Calderon M, Andersen PS, Shamji M, Durham SR. Protocol for a randomised, double-blind, placebo-controlled study of grass allergen immunotherapy tablet for seasonal allergic rhinitis: time course of nasal, cutaneous and immunological outcomes. Clin Transl Allergy. 2015 Dec 17;5:43. doi: 10.1186/s13601-015-0087-2. eCollection 2015. PMID 26682038

RESULTS

PARTICIPANT FLOW:
Groups:
- Grazax: The active treatment arm received active grass pollen immunotherapy tablet (AIT), Grazax Oral Lyophilisate 75,000 standardised quality units tablet (SQ-T) once daily.
  Grazax: The active treatment arm will receive active grass pollen immunotherapy tablet (AIT), Grazax Oral Lyophilisate 75,000 SQ-T once daily.
- Grazax Placebo: This arm received Grazax placebo once daily which contains the same composition as in the active Grazax tablet with the only difference being the exclusion of the grass pollen allergen extract.
  Grazax Placebo: This arm will receive Grazax placebo once daily which contains the same composition as in the active Grazax tablet with the only difference being the exclusion of the grass pollen allergen extract.
Period: Overall Study
Arm/Group | Grazax | Grazax Placebo
Started | 23 | 23
Completed | 21 | 19
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Grazax: The active treatment arm received active grass pollen immunotherapy tablet, Grazax Oral Lyophilisate 75,000 standardised quality units tablet once daily.
- Grazax Placebo: This arm received Grazax placebo once daily which contains the same composition as in the active Grazax tablet with the only difference being the exclusion of the grass pollen allergen extract.
- Total: Total of all reporting groups
Arm/Group | Grazax | Grazax Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Median (Standard Deviation); unit: years] | 31.5 (2.12) | 36.9 (1.97) | 34.2 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 13 | 18 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23 | 23 | 46
Specific Immunoglobulin E (IgE) [Median (Standard Deviation); unit: kU/l] | 14.4 (3.12) | 14.17 (2.81) | 14.28 (2.96)

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Symptom Score After Nasal Allergen Challenge (NAC)
Description: The total nasal symptom score at one hour after grass pollen nasal allergen challenge in active versus placebo treated participants after treatment period. Score ranges from minimum 0 point to maximum of 12 points. Higher score is more severe symptoms.
Time Frame: 60 minutes post-challenge after 12 months of treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Grazax | Grazax Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | 3.37 [2.7 to 4.05] | 4.71 [4 to 5.4]
Statistical Analysis 1: Comparison: Grazax vs Grazax Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided — calculated

2. Secondary Outcome: Early Phase Intradermal Test
Description: Mean Diameter in millimetre of EPR skin responses to intradermal grass pollen allergen injection at 12 months in active versus placebo treated participants. The larger the diameter the worst symptoms.
Time Frame: after 12 months of treatment
Measure: Mean (Standard Error); unit: Millimiters
Arm/Group | Grazax | Grazax Placebo
Number analyzed (Participants) | 23 | 23
Millimiters | 15.3 (1.1) | 20.2 (1.1)

3. Secondary Outcome: Late Phase Intradermal Test
Description: Mean Diameter in millimetre of LPR skin responses to intradermal grass pollen allergen injection at 12 months in active versus placebo treated participants. The larger the diameter the worst symptoms
Time Frame: after 12 months of treatment
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Grazax | Grazax Placebo
Number analyzed (Participants) | 23 | 23
millimeters | 52.6 (3.4) | 74.6 (3.4)

4. Secondary Outcome: Change From Baseline in Delta Peak Nasal Inspiratory Flow in L/Min
Description: Nasal patency assessed at 60 minutes after nasal allergen challenge 12 months after treatment. The lower the peak nasal inspiratory flow the blockage nasal patency is.
Time Frame: 60 minutes post-challenge after 12 months of treatment
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Grazax | Grazax Placebo
Number analyzed (Participants) | 23 | 23
L/min | -29.2 [-44.8 to -13.5] | -72.5 [-88.8 to -56.1]
Statistical Analysis 1: Comparison: Grazax vs Grazax Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided

5. Secondary Outcome: End of Season Global Rhinitis Symptoms
Description: Hayfever symptoms during last pollen season after start of treatment. Score on a scale ranges from minimum 0 point to maximum of 100 points. Higher score is more severe symptoms.
Time Frame: after treatment at 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Grazax | Grazax Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | 40.4 (5.18) | 54.97 (5.43)
Statistical Analysis 1: Comparison: Grazax vs Grazax Placebo; Null Hypothesis was no difference between Grazax and Placebo treatment at 12 months. 80% power to detect 30% difference in total nasal symptom score (TNSS) after nasal challenge; Test type: Superiority; Comparison of nasal symptom score at 0-60 mins after nasal challenge after 12 months treatment with Grazax compared to Placebo treatment. Mixed model analysis. 80% power to detect a 30% difference at p<0.05

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Grazax | Grazax Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 22/23 | 20/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazax (N=23) | Grazax Placebo (N=23)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Allergic Reaction (Immune system disorders) | 19 (23) | 3 (3)
Tooth ache (General disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Common cold/URTI (Infections and infestations) | 15 (88) | 20 (60) — Upper respiratory tract infection
Headache (Nervous system disorders) | 5 (38) | 5 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT02005627/SAP_000.pdf
  • Study Protocol (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02005627/Prot_001.pdf
  • Informed Consent Form (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02005627/ICF_002.pdf